CLINICAL TRIAL: NCT06257745
Title: Evaluation of the Revised Enhanced Recovery After Cardiac Surgery Protocol. A Prospective Audit.
Brief Title: Audit of the Revised PACU Centric ERACS Program
Acronym: ERACS2
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s68333
Record Dates: First submitted 2024-01-25; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-01

CONDITIONS: Enhanced Recovery After Surgery; Cardiac Surgical Procedures
MeSH Terms: interventions — Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ERACS group: Any patient admitted to our post-anesthesia care unit following cardiac surgery and planned for overnight stay.
  Interventions: Other: Compliance with ERACS guideline as described in the current ERACS guidelines from Engelman et al. 2019

INTERVENTIONS:
Other: Compliance with ERACS guideline as described in the current ERACS guidelines from Engelman et al. 2019 — Compliance with the interventions as proposed in the ERACS guidelines and described in our previous publication (https://doi.org/10.1016/j.jtcvs.2022.07.010

SUMMARY:
A previous audit (S63843) found an association between improved compliance with these interventions and postoperative outcomes (hospital length of stay (LOS) and presence of ≥1 postoperative complication). The investigators found that every 10% increase in compliance was associated with an increased risk (HR=1.25, p=0.0008) for early discharge. In addition, improved compliance was also associated with a reduction (OR=0.60, p=0.0003) of postoperative complications. Based on these findings, improving compliance with current guidelines remains a hurdle that clinicians should overcome. The investigators previous retrospective study was unable to identify the reason for non-compliance and the relation to postoperative outcomes. Therefore, a prospective audit is warranted to assess reach, fidelity, and dose of the different interventions.

DETAILED DESCRIPTION:
Trial Design:

Prospective audit in patients undergoing cardiac surgery and planned for overnight stay within our post-anesthesia care unit (PACU) enhanced recovery after cardiac surgery (ERACS) program. The medical records of all patients will be evaluated for the implementation of various interventions of our ERACS program (primary objective). For the secondary objective the investigators will assess the occurrence of postoperative complications and hospital LOS.

For benchmarking (third objective), the investigators will compare the findings with the results of a previous audit (S63843).(4) Data in this retrospective audit was collected from the electronic patient registry (KWS = Klinisch Werk Station). This included all interventions described in the ERACS guidelines. In addition, postoperative complications that occurred up to 7 days were also collected.

Data management:

Data will be obtained, according to the strategy used in the previous audit (S63843), by a research collaborator and an anesthesiologist using the medical records of the included patients. Appropriate data will also be collected from the preoperative anesthesia evaluation sheets (digitally stored in the hospital information system, KWS Nexus health) and from all intra- and postoperative anesthesia records up to 30 days after the index surgery.

Statistics:

The investigators aim for a convenience sample of 1-year recruitment, from January 1st 2024 until December 31st 2024 and expect to include approximately 350 cardiac surgical patients in this ERACS audit.

Patient characteristics will be tabulated as absolute numbers, percentages, mean and standard deviation, Objective 1 95% confidence intervals will be reported for the mean (or median) percentage compliances well as for each of the interventions separately, the proportion of patients who adhere to the intervention.

Objective 2 Logistic regressions will be used to verify the relation between the percentage adherence and the presence of a complication (for each complication separately and for the composite endpoint). Odds ratios and 95% confidence intervals will be reported. These analyses will also be performed for the adherence at each intervention separately (fidelity and dose). Spearman correlations and MWU tests will be used to explore relations between adherence (percentage and each intervention separately) and length of hospital stay. Given the possible presence of in-hospital mortality, a LOS value higher than the maximal observed value of the discharged patients will be given to patients who die in the hospital when applying these rank-based methods. Further, Cox regressions will be used to model the cause-specific hazard in presence of in-hospital mortality and hazard ratios (with 95%CI) will be given. A multivariable logistic regression will be used to verify if the relation between protocol adherence and postoperative complications is not confounded by patient (e.g. EuroSCORE II) and procedural (e.g. type of surgery being valvular, bypass or minimally invasive) characteristics. To verify the independent impact of protocol adherence on length of stay, a multivariable Cox regression will be used.

Objective 3 For benchmarking purposes, the percentage adherence will be compared between current sample and the data of the retrospective study using a linear normal model, correcting for potential differences in patient-mix (patient and procedural characteristics) between both periods. Note however that differences are expected to be minimal, since the same inclusion criteria were used, and the accrual period covered a full year. To compare the adherence to each intervention separately and to compare the complication rate(s) a logistic regression will be used.

A p-value of less than 0.05 will be considered statistically significant. Given the large number of planned statistical tests, a single significant p-value will be interpreted with caution.

ELIGIBILITY:
Inclusion Criteria:

* Included in our post anesthesia care unit centric ERACS program during 2024

Exclusion Criteria:

* Patients transferred to the PACU but awaiting planned admission to the intensive care unit following cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any patient undergoing cardiac surgery in our hospital and requiring admittance to a high-depency unit for overnight stay.
Sampling Method: Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Overall percentage of compliance with the 24 interventions of the ERACS guidelines | From 6 week prior to surgery up to 1 month after surgery
  Performed interventions as described in the ERACS guidelines and adapted to local standards

SECONDARY OUTCOMES:
Hospital length of stay following the index surgery | From date of surgery until the date of hospital discharge or date of death from any cause, whichever came first, assessed up to 30days.
  Number of nights in the hospital
Occurrence of each postoperative complication during the first 7 days | From date of surgery up to 7 postoperative days
  Complications as described in our previous publication (https://doi.org/10.1016/j.jtcvs.2022.07.010)
Composite endpoint of 1 or more postoperative complications | From date of surgery up to 7 postoperative days
  Complications as described in our previous publication (https://doi.org/10.1016/j.jtcvs.2022.07.010)
Percentage of patients in whom each ERACS intervention was performed as intended (referred to as fidelity) | From 6 week prior to surgery up to 1 month after surgery
  Interventions as described in the ERACS guidelines
Percentage of patients in whom each the frequency of ERACS intervention was performed as planned (referred to as dose) | From 6 week prior to surgery up to 1 month after surgery
  Number of interventions as described in the ERACS guidelines

OTHER OUTCOMES:
Benchmarking purpose | From 6 week prior to surgery up to 1 month after surgery
  the percentage adherence will be compared between current sample and the data of the retrospective study using a linear normal model, correcting for potential differences in patient-mix (patient and procedural characteristics) between both periods. Note however that differences are expected to be minimal, since the same inclusion criteria were used, and the accrual period covered a full year. To compare the adherence to each intervention separately and to compare the complication rate(s) a logistic regression will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Danny Feike Hoogma, MD, PhD, Principal Investigator — Anesthesiology
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
IPD is available upon request from the primary investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available following the publication of the current audit in a peer reviewed journal
Access Criteria: Detailes request for IPD needs to be addressed to the PI.

REFERENCES:
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Background] Hoogma DF, Croonen R, Al Tmimi L, Tournoy J, Verbrugghe P, Fieuws S, Rex S. Association between improved compliance with enhanced recovery after cardiac surgery guidelines and postoperative outcomes: A retrospective study. J Thorac Cardiovasc Surg. 2024 Apr;167(4):1363-1371.e2. doi: 10.1016/j.jtcvs.2022.07.010. Epub 2022 Jul 19. PMID 35989120
- [Background] Fleming IO, Garratt C, Guha R, Desai J, Chaubey S, Wang Y, Leonard S, Kunst G. Aggregation of Marginal Gains in Cardiac Surgery: Feasibility of a Perioperative Care Bundle for Enhanced Recovery in Cardiac Surgical Patients. J Cardiothorac Vasc Anesth. 2016 Jun;30(3):665-70. doi: 10.1053/j.jvca.2016.01.017. Epub 2016 Jan 16. PMID 27321791
- [Background] Van Grootven B, Jeuris A, Jonckers M, Devriendt E, Dierckx de Casterle B, Dubois C, Fagard K, Herregods MC, Hornikx M, Meuris B, Rex S, Tournoy J, Milisen K, Flamaing J, Deschodt M. How to implement geriatric co-management in your hospital? Insights from the G-COACH feasibility study. BMC Geriatr. 2022 May 2;22(1):386. doi: 10.1186/s12877-022-03051-1. PMID 35501840